CLINICAL TRIAL: NCT06391138
Title: The Effect of Obstructive Sleep Apnea on Pregnancy and Fetal Outcomes
Brief Title: The Effect of OSA on Pregnancy and Fetal Outcomes
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Xiaowan Du, Principal Investigator, Peking University First Hospital
Other Study IDs: PKUFH ENT OSAP V1.0
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Pregnancy; Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Continuous Positive Airway Pressure — The intervention in this study involves the use of Continuous Positive Airway Pressure (CPAP) treatment. CPAP is a commonly used therapy for obstructive sleep apnea (OSA) and other sleep-related breathing disorders. The principle of CPAP treatment lies in maintaining a constant airway pressure during sleep to prevent the collapse of the upper airway and ensure unobstructed breathing. The patient wears a mask connected to a CPAP machine, which generates a steady stream of air to provide the necessary pressure.

SUMMARY:
This cohort study aims to investigate the impact of obstructive sleep apnea hypopnea syndrome (OSA) on pregnancy and fetal outcomes. The hypothesis posits that OSA may aggravate pregnancy complications, elevate the risk of adverse pregnancy outcomes, and potentially impact fetal development.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with a confirmed diagnosis of OSA based on polysomnography or other validated sleep monitoring techniques.
* Pregnant women who are willing to participate in the study and provide informed consent.

Exclusion Criteria:

* Pregnant women with other respiratory or sleep disorders that may confound the diagnosis of OSA.
* Pregnant women with severe comorbidities or medical conditions that may significantly impact pregnancy outcomes.
* Pregnant women who have undergone surgical treatment for chronic tonsillitis or OSA during the study period.
* Pregnant women who refuse to participate in the study or are unable to provide informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnancy
Study Population: Pregnant women with OSA who have established prenatal care records and undergone antenatal check-ups at PKUFH
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
rate of pre-eclampsia/ eclampsia | 10 months

SECONDARY OUTCOMES:
rate of preterm birth | 10 months

OTHER OUTCOMES:
birth weight | 10 months
  birth weight of newborns measured in grams
length of newborns | 10 months
  length of newborns measured in centimeters
The Apgar score of newborns | 10 months
  The Apgar score consists of five main indicators: skin color, heart rate, response to stimulation, muscle tone, and respiration. Each indicator is scored from 0 to 2, with a total score of 10. This scoring method serves as a guiding tool for the resuscitation of newborns with asphyxia and could provide a degree of predictive value for the neurological development of infants in the future.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaowan Du, Study Director — Peking University First Hospital

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be provided upon request.